CLINICAL TRIAL: NCT00136331
Title: Phase Ia Study of a Pandemic Influenza Vaccine
Brief Title: Study of a Pandemic Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Dr Russell Basser, CSL Limited
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CSLCT-PAN-05-12
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2008-11

CONDITIONS: Influenza
Keywords: Pandemic; Influenza; Prevention; Vaccine; Prevention of Pandemic Influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Pandemic influenza vaccine

SUMMARY:
The World Health Organisation has warned that an influenza pandemic is inevitable. The avian influenza H5N1 virus strain is the leading candidate to cause the next avian influenza pandemic. This study will test the safety and immunogenicity of a H5N1 pandemic influenza vaccine in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* History of Guillain-Barre syndrome or active neurological disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400
Dates: Start 2005-10; Study Completion 2006-11

PRIMARY OUTCOMES:
Safety and immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Terry M Nolan, Principal Investigator — Murdoch Childrens Research Institute
Locations (2):
- Australia (2):
  - CMAX, a division of IDT Australia, Adelaide, South Australia
  - Murdoch Childrens Research Institute, Melbourne, Victoria

REFERENCES:
- [Derived] Nolan TM, Richmond PC, Skeljo MV, Pearce G, Hartel G, Formica NT, Hoschler K, Bennet J, Ryan D, Papanaoum K, Basser RL, Zambon MC. Phase I and II randomised trials of the safety and immunogenicity of a prototype adjuvanted inactivated split-virus influenza A (H5N1) vaccine in healthy adults. Vaccine. 2008 Aug 5;26(33):4160-7. doi: 10.1016/j.vaccine.2008.05.077. Epub 2008 Jun 13. PMID 18599164